CLINICAL TRIAL: NCT05240833
Title: VExUS-guided Fluid Management in Patients With Acute Kidney Injury in the Intensive Care Unit
Acronym: AKIVEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0487
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Acute; Kidney; Disease, Acute; Critical Illness; Volume Overload; Fluid Overload
MeSH Terms: conditions — Acute Kidney Injury; Disease; Critical Illness; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VExUS-Guided Arm (Experimental): VExUS results will be available for the treating physician. Patients will be treated according to current clinical practice. The use of diuretic and diuretic dosage will depend on treating physician's criteria.
  Interventions: Diagnostic Test: VExUS Score

INTERVENTIONS:
Diagnostic Test: VExUS Score — The VExUS-Guided Arm care team will be informed of the Day 0 VExUS immediately after the ultrasound is performed and given a suggested target for the following 48 hours as follows:
  * VExUS 0: There is no evidence of venous congestion.
  * VExUS 1: There is evidence of mild venous congestion. The investigators recommend targeting a net neutral or negative fluid balance with diuresis.
  * VExUS 2-3: There is evidence of moderate to severe venous congestion. The investigators recommend targeting a fluid balance of negative 1-2L with diuresis.
  * If the investigator cannot obtain ultrasound images of sufficient quality to calculate VExUS, the care team will be informed that there is no recommendation for that subject on that day.

SUMMARY:
A quasi experimental study that aims to verify whether the incorporation of VExUS in patients with AKI in the Intensive Care Unit (ICU) may prompt tailored interventions to increases the number of days free from Renal Replacement Therapy (RRT) during the first 28 days.

DETAILED DESCRIPTION:
Fluid overload is associated with organ dysfunction, such as Acute Kidney Injury (AKI), and increased mortality. It remains unclear if fluid overload is merely an epiphenomenon in critically ill patients or if organ congestion is a mediator of complications. Considering AKI related to fluid overload, diuretic therapy would reduce venous congestion and improve renal blood flow. The Venous Excess Ultrasound score (VExUS) identifies clinically significant venous congestion and indicates a high risk of post-operative AKI. This quasi-experimental study aims to verify whether the incorporation of VExUS in patients with AKI in the Intensive Care Unit (ICU) may prompt tailored interventions to increases the number of days free from Renal Replacement Therapy (RRT) during the first 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Non-elective ICU admission
* Severe acute kidney injury (AKI) defined either: A ≥ 2-fold increase in serum creatinine from a known pre-morbid baseline or during the current hospitalization OR Urine output < 6.0 mL/kg over the preceding 12 hours

Exclusion Criteria:

* Life-threatening indication of RRT (defined as intractable hyperkalaemia, acidosis, uraemic symptoms) at Day 0
* RRT before recruitment
* Use of Extracorporeal membrane oxygenation (ECMO)
* Hepatic cirrhosis or other condition with portal hypertension
* Lack of commitment to provide RRT as part of limitation of ongoing life support
* Known pre-hospitalization advanced chronic kidney disease, defined by an estimated glomerular filtration rate < 30 mL/min/1.73 m2 or chronic RRT
* Refusal to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Renal replacement therapy | Day 28
  Number of days free from renal replacement therapy during the first 28 days

SECONDARY OUTCOMES:
Mortality | Day 28
KDIGO category for AKI | 48 hours
  Variation in Kidney Disease: Improving Global Outcomes (KDIGO) criteria for AKI after 48 hours. Reducing the KDIGO category is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: MARCIO M BONIATTI, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No